CLINICAL TRIAL: NCT00002668
Title: PATIENT SKILLS FOR CANCER PAIN CONTROL IN PATIENTS WITH METASTATIC BREAST OR PROSTATE CANCER
Brief Title: Pain Control in Patients With Recurrent or Metastatic Breast or Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDR0000064257; U10CA021115 (NIH); ECOG-3Z93; NCI-P95-0068
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Pain; Prostate Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV prostate cancer; recurrent prostate cancer; pain
MeSH Terms: conditions — Breast Neoplasms; Pain; Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (Active Comparator): Standard pain management interventions usually given by hospital staff
  Interventions: Behavioral: Observation
- Educational Intervention and Behavioral Skills Training (Experimental): Patients participated in a program including video presentations, written materials, and coaching in behavioral skills to improve pain control (not to reduce analgesic use).
  Interventions: Behavioral: Educational Intervention and Behavioral Skills Training

INTERVENTIONS:
Behavioral: Observation
  Arms: Observation
Behavioral: Educational Intervention and Behavioral Skills Training
  Arms: Educational Intervention and Behavioral Skills Training

SUMMARY:
RATIONALE: An outpatient educational and behavioral skills training program may help patients with metastatic breast or prostate cancer live longer and more comfortably.

PURPOSE: This randomized clinical trial studies whether an outpatient educational and behavioral skills training program will improve pain control in patients who have metastatic or recurrent breast or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the feasibility of implementing an outpatient education and behavioral skills training program for pain control in a multi-institution setting.
* Evaluate whether patient education and behavioral skills training improve cancer pain control in patients with recurrent or metastatic breast or prostate cancer.
* Amend the protocol, with the approval of the Division of Cancer Prevention and Control, to a groupwide 3-arm study if analysis demonstrates feasibility and potential efficacy of the patient education and behavioral skills training program.

OUTLINE: This is a randomized study. Patients are stratified according to diagnosis (breast vs prostate cancer), initial "pain worst" score (4-6 vs 7 or higher), and participating institution. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive standard pain management.
* Arm II: Patients receive educational intervention (booklets, audiotapes, and videotapes) and behavioral skills training (including a schedule of practice relaxation sessions) in addition to standard pain management. Patients receive a follow-up phone call within 48-72 hours of intervention to review pain status.

Patients on both arms undergo pain and psychological assessments on days 1 and 15.

PROJECTED ACCRUAL: A total of 96 patients (48 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Recurrent or metastatic breast or prostate cancer
* "Pain worst" score of 4 or greater on the Brief Pain Inventory
* No prior enrollment on this study (patients treated during the run-in period are ineligible for randomization)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No major psychiatric illness, including the following DSM-III-R diagnoses:

  * Bipolar disorder
  * Schizophrenia
  * Major depression
  * Multiple personality disorder
  * Psychotic disorder
  * Dementia
  * Outpatient status required

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 28 days since prior palliative radiotherapy to major site(s) of pain

Surgery:

* Greater than 30 days since prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1996-02-14 (Actual); Primary Completion 1998-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Change in pain assessed using the Brief Pain Inventory | Assessed over 15 days
  Change in worst pain from baseline to day 15

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cleeland, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (18):
- United States (15):
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico